CLINICAL TRIAL: NCT04983914
Title: Retrospective Non-Interventional Study to Evaluate the Patient Benefit of Transcorneal Electrostimulation (TES)
Brief Title: Retrospective NIS to Evaluate the Patient Benefit of TES
Status: Completed | Type: Observational
Sponsor: Okuvision GmbH (Industry)
Collaborators: CONET GmbH - Clinical Operations Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: TES-NIS2021
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Retinitis Pigmentosa
Keywords: Transcorneal Electrostimulation; TcES; TES; Inherited retinal dystrophy; Retinopathia pigmentosa; Retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcorneal Electrostimulation via OkuStim System — Transcorneal electrostimulation, usually applied once per week for 30 min (home-use).
  Other Names: TcES; TES; OkuStim

SUMMARY:
In this retrospective non-interventional study (NIS), the subjective and objective benefit of patients with retinitis pigmentosa (and other dystrophies like Usher, Choroideremia or cone-rod dystrophy), who have been prescribed the therapy of transcorneal electrostimulation (TcES) with the OkuStim System, is assessed.

DETAILED DESCRIPTION:
The medical device OkuStim received the CE mark (a symbol of free marketability in the European Economic Area) in 2011 and is commercially available for patients in Europe since 2014. Since then, patients with retinitis pigmentosa and other dystrophies have regularly applied the therapy of transcorneal electrostimulation (TcES) with OkuStim. So far, the benefits of the therapy and the experiences of the patients with regular, multi-year use have not been systematically recorded.

In this retrospective non-interventional study (NIS) with patients which have been using TcES since >1 year, data present for visual field, best-corrected visual acuity (BCVA) and central foveal thickness (as assessed via OCT) is collected. In addition, reasons for discontinuation of therapy and patient satisfaction with TcES are assessed via a questionnaire. Side-effects are also recorded, if present in the patient files.

ELIGIBILITY:
Inclusion Criteria:

* Use of TcES for >1year
* Willing and able to consent

Exclusion Criteria:

* Not willing and able to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been prescribed the OkuStim System and who use the therapy for more than one year are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Visual field | Baseline and then all data present in patient files after begin of therapy. Depending on how long the patient already uses OkuStim, the time frame varies between 1 year and several years after commencement of therapy.
  Assessment of changes compared to baseline (before TcES was started)

SECONDARY OUTCOMES:
Best-corrected visual acuity | Baseline and then all data present in patient files after begin of therapy. Depending on how long the patient already uses OkuStim, the time frame varies between 1 year and several years after commencement of therapy.
  Assessment of changes compared to baseline (before TcES was started)
Central foveal thickness | Baseline and then all data present in patient files after begin of therapy. Depending on how long the patient already uses OkuStim, the time frame varies between 1 year and several years after commencement of therapy.
  Assessment of changes compared to baseline (before TcES was started)

OTHER OUTCOMES:
Reasons for discontinuation of therapy and patient satisfaction | Patients are asked to fill out the questionnaire once. Depending on how long the patient already uses OkuStim, the time frame varies between 1 year and several years after commencement of therapy
  Custom-made questionnaire to assess reasons for discontinuation of therapy and patient satisfaction
Adverse events | All data present in patient files after begin of therapy. Depending on how long the patient already uses OkuStim, the time frame varies between 1 year and several years after commencement of therapy.
  Adverse events will be recorded if present in the patient files. Only device-related adverse events will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Scholl, Prof. Dr., Principal Investigator — Department of Ophthalmology, University of Basel, Switzerland; Katarina Stingl, Prof. Dr., Principal Investigator — University Eye Hospital Tuebingen, Tuebingen, Germany
Locations (4):
- Germany (3):
  - Universitätsklinikum Heidelberg, Augenklinik, Heidelberg
  - Klinikum Stuttgart gKAöR, Augenklinik Standort Mitte (Katharinenhospital), Stuttgart
  - Universitäts-Augenklinik Tübingen, Abt. für Augenheilkunde, Tübingen
- Universitätsspital Basel, Augenklinik, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zabek O, Camenzind Zuche H, Muller U, Scholl HPN, Rickmann A, Della Volpe Waizel M. Optical coherence tomography angiography findings in patients undergoing transcorneal electrical stimulation for treating retinitis pigmentosa. Graefes Arch Clin Exp Ophthalmol. 2021 May;259(5):1167-1177. doi: 10.1007/s00417-020-04963-7. Epub 2020 Oct 10. PMID 33037922
- [Background] Jolly JK, Wagner SK, Martus P, MacLaren RE, Wilhelm B, Webster AR, Downes SM, Charbel Issa P, Kellner U, Jagle H, Ruther K, Bertelsen M, Bragadottir R, Prener Holtan J, van den Born LI, Sodi A, Virgili G, Gosheva M, Pach J, Zundorf I, Zrenner E, Gekeler F. Transcorneal Electrical Stimulation for the Treatment of Retinitis Pigmentosa: A Multicenter Safety Study of the OkuStim(R) System (TESOLA-Study). Ophthalmic Res. 2020;63(3):234-243. doi: 10.1159/000505001. Epub 2019 Nov 26. PMID 31775146
- [Background] Schatz A, Pach J, Gosheva M, Naycheva L, Willmann G, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Messias A, Gekeler F. Transcorneal Electrical Stimulation for Patients With Retinitis Pigmentosa: A Prospective, Randomized, Sham-Controlled Follow-up Study Over 1 Year. Invest Ophthalmol Vis Sci. 2017 Jan 1;58(1):257-269. doi: 10.1167/iovs.16-19906. PMID 28114587
- [Background] Schatz A, Rock T, Naycheva L, Willmann G, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Messias A, Gekeler F. Transcorneal electrical stimulation for patients with retinitis pigmentosa: a prospective, randomized, sham-controlled exploratory study. Invest Ophthalmol Vis Sci. 2011 Jun 23;52(7):4485-96. doi: 10.1167/iovs.10-6932. PMID 21467183
- [Background] Sinim Kahraman N, Oner A. Effect of Transcorneal Electrical Stimulation on Patients with Retinitis Pigmentosa. J Ocul Pharmacol Ther. 2020 Oct;36(8):609-617. doi: 10.1089/jop.2020.0017. Epub 2020 May 19. PMID 32429728
- [Background] Della Volpe-Waizel M, Zuche HC, Muller U, Rickmann A, Scholl HPN, Todorova MG. Metabolic monitoring of transcorneal electrical stimulation in retinitis pigmentosa. Graefes Arch Clin Exp Ophthalmol. 2020 Jan;258(1):79-87. doi: 10.1007/s00417-019-04522-9. Epub 2019 Nov 12. PMID 31713752